CLINICAL TRIAL: NCT06988943
Title: Construction and Evaluation of a Hospital-Community Health Collaboration Model Empowered by Digital Technology for Lung Cancer Screening
Brief Title: Early Intervention Strategies for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Director, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ES-2024-193-01-001
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Lung Neoplasms
Keywords: Screning test; Lung cancer; LDCT; Low-dose CT
MeSH Terms: conditions — Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digitally enabled low-dose CT screening Group (Experimental)
  Interventions: Device: Low-dose CT screening; Device: AI full-lung model interpretation system; Device: Digital Health Platform

INTERVENTIONS:
Device: Low-dose CT screening — Low-dose CT screening is conducted at primary healthcare institutions, and patients with detected lung nodules are referred to hospitals for further examination
Device: AI full-lung model interpretation system — Using artificial intelligence technology to assist in the interpretation of CT images
Device: Digital Health Platform — Community health centers and streets in Guangzhou use a program called "Fei Anxin" to manage residents' information in a unified way

SUMMARY:
Low-dose CT (LDCT）can detect and treat lung cancer earlier and more quickly, while expanded screening coverage helps reduce the incidence and mortality of respiratory diseases such as lung cancer. This study aims to conduct a single-arm cluster randomized trial of digitally enabled LDCT in Guangzhou to assess its intervention effectiveness and cost-effectiveness.

DETAILED DESCRIPTION:
This study uses a single-arm design to assign community health service centers in two districts of Guangzhou (Liwan and Baiyun) to the intervention group. A historical self-comparison design is employed. The intervention measures utilize a digital empowerment model for lung cancer screening, which includes the following components: ① Digital health platform: Each street and community health center manages resident information through the Lung Health mini-program; ② AI-based full-lung model reading system: Using artificial intelligence technology to assist in interpreting CT images; ③ Low-dose CT screening: Low-dose CT screening is conducted at primary healthcare institutions, and patients with detected lung nodules are referred to hospitals for further examination. The sampling method used is Probability Proportional to Size (PPS), with an expected sample size of 16000. Participants will complete the "Lung Cancer Health Questionnaire" to collect individual-level confounding factors. Screening data will be collected through the "Fei'anxin" mini-program, and diagnostic data will be provided by designated hospitals and the First Affiliated Hospital of Guangzhou Medical University. The primary outcome of the study is the proportion of early-stage lung cancer in the screening population, defined as the number of early-stage lung cancer cases divided by the total number of people screened. An economic evaluation of the lung cancer CT screening will also be conducted.

ELIGIBILITY:
1.Community Health Service Centers (Cluster Level)

1. Inclusion Criteria The community health service center must be located within one of the 11 districts of Guangzhou.

   The center must manage a population of over 10,000 elderly individuals. The center should be equipped with at least one CT machine and have qualified medical personnel, such as radiologists, radiologic technicians, and nursing staff.
2. Exclusion Criteria Community health centers currently participating in other public health projects or studies that may affect screening results.

Community health service centers where researchers cannot collect data or conduct follow-up.

2. Screening Subjects (Individual Level)

1. Inclusion Criteria Aged 40-75 years. Residing in the community participating in the study for a long time. No known history of lung cancer and has not undergone lung cancer screening in the past three months.

   Able to understand and willing to sign the informed consent form, and able to participate in long-term follow-up.
2. Exclusion Criteria Individuals diagnosed with lung cancer. Individuals with severe other health issues that make them unsuitable for CT imaging.

Individuals unable to understand the study protocol or who cannot provide informed consent due to cognitive impairments.

Individuals participating in other clinical trials that may affect the results of this study.

Individuals unable to undergo follow-up.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The early diagnosis rate of lung cancer | Within 1 year after the intervention is implemented

SECONDARY OUTCOMES:
The number of participants in lung cancer screening | Within 1 year after the intervention is implemented
Number of individuals with positive screening results | Within one year after the intervention is implemented
3-month follow-up rate. | Within three months after the intervention is implemented
One-year follow-up rate | Within 1 year after the intervention is implemented
Diagnosis rate | Within 1 year after the intervention is implemented
False positive rate for nodules | Within 1 year after the intervention is implemented
Positive predictive value for nodules | Within 1 year after the intervention is implemented
Average time to read CT images | Within 1 year after the intervention is implemented
CT screening complications | Within 1 year after the intervention is implemented
Complications of diagnostic tests | Within 1 year after the intervention is implemented

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No